CLINICAL TRIAL: NCT06595745
Title: Testing a Combined Approach to Control Mosquito-Borne Diseases At Scale
Brief Title: Testing Combined IIT-SIT to Control Mosquito-Borne Diseases At Scale
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Universidad Autónoma de Yucatán (Other); Emory University (Other)
Responsible Party: Principal Investigator, Zhiyong Xi, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00010509; 7200AA23FA00021 (Other: USAID)
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dengue; Zika; Chikungunya
Keywords: Wolbachia; IIT; SIT; Aedes aegypti; Dengue; Zika; Chikungunya
MeSH Terms: conditions — Dengue; Zika Virus Infection; Chikungunya Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Release sites (Experimental): Traditional mosquito control will be applied, followed by weekly release of Wolbachia wAlbB-infected Aedes aegypti males to induce sterile mating with wild female mosquitoes.
  Interventions: Genetic: Wolbachia induced incompatible mating; Combination Product: Standard traditional chemical mosquito control
- Control sites with traditional mosquito control only (Active Comparator): Traditional mosquito control will be applied but no mosquito release will occur in the control sites
  Interventions: Combination Product: Standard traditional chemical mosquito control

INTERVENTIONS:
Genetic: Wolbachia induced incompatible mating — The intervention will be performed by weekly release of male Aedes aegypti carrying Wolbachia (wAlbB strain) to mate with wild females, resulting in the death of their eggs for birth control. Before release, these males will be irradiated with X-rays to minimize the chance of any residual fertile female releases. The intervention will lead to Ae. aegypti population suppression or even elimination and preventing dengue transmission in release sites.
  Other Names: Incompatible insect technique; Sterile insect technique
  Arms: Release sites
Combination Product: Standard traditional chemical mosquito control — Traditional and commonly used chemical insecticide will be applied to reduce the mosquito population

SUMMARY:
Mosquito-borne diseases cause suffering for hundreds of millions of people and claim more than 700,000 lives yearly. Diseases such as dengue, Zika, and chikungunya cause symptoms similar to malaria and are endemic in many parts of the world, yet there are no treatments for them nor vaccines for Zika and chikungunya. Mosquito control, particularly of the Aedes aegypti species, is seen as a potentially effective solution to slow or stop the spread of these diseases but has not yet demonstrated significant, sustainable impacts on disease transmission. The investigators will aim to significantly control or eliminate local foci (hot-spots) of dengue, chikungunya and Zika transmission and significantly reduce disease transmission by implementing a combined incompatible and sterile insect technique (IIT-SIT) program based on the release of male Aedes aegypti carrying Wolbachia (wAlbB strain) that have been previously irradiated with X-rays (to minimize the chance of fertile female releases). The investigators will implement a two-arm cluster randomized controlled trial to evaluate the epidemiological and entomological impact of population suppression via IIT-SIT on Aedes-borne diseases in the city of Merida, Mexico. Primary endpoint of the trial is the incidence of laboratory Aedes-borne viruses detected by the passive surveillance system of Mexico. Secondary endpoints will allow estimating the level of suppression of Ae. aegypti populations. This trial design will allow establishing a link between epidemiologic, entomo-virological and entomological indicators to determine the effectiveness of IIT-SIT in real world conditions. The approach is novel because it effectively eliminate vectors, such as urban, outdoor, daytime biting mosquitoes, which are not susceptible to standard vector control approaches, by targeting cryptic and inaccessible mosquito habitats. In addition, the intervention has the below advantages comparing to existing alternatives: (i) highly competitive males are used for release as Wolbachia-infected males have the mating competitiveness equal to wild-type males; (ii) release can continue until population elimination is reached as a low dose of radiation is used to sterilize females for preventing risk of population replacement; (iii) any residual females contaminated in released male pools is resistant to pathogens; (iv) public acceptance of release of Wolbachia-infected males can be easily achieved, because Wolbachia are bacteria naturally presenting in ~50 percent of insect species, and male mosquitoes neither bite nor transmit diseases and can be self-limiting post release; (v) it will not impact non-target species. Successful findings from this study will pave the way for future expansions of the combined IIT-SIT to the entire city and nationwide using a rolling-carpet strategy, which has been successfully demonstrated for area-wide control of screwworm and medfly in Latin America.

ELIGIBILITY:
Inclusion Criteria:

* All residents in the release sites will be included in the studies

Exclusion Criteria:

* No exclusion will be performed.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15243 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Epidemiological impact of combined IIT-SIT | Up to 19 months
  Incidence of symptomatic Aedes-borne virus (dengue, chikungunya, Zika) confirmed by laboratory testing by the Yucatan Ministry of Health.

SECONDARY OUTCOMES:
Entomological impact of combined IIT-SIT | Up to 19 months
  Number of Aedes aegypti females infected with dengue, chikungunya or Zika virus (quantified as minimum infection rate, MIR); Number of Aedes aegypti females collected indoors (during 10-minute collections) using Prokopack aspirators; Number of Aedes aegypti females collected in the peridomicile with BG-sentinel traps.

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Vazquez Professor Prokopec, PhD, Study Chair — Emory University
Locations (1):
- Laboratorio para el Control Biolo´gico de Aedes aegypti (LCB-UADY), Universidad Autónoma de Yucatán, Mérida, Yucatán, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liang X, Tan CH, Sun Q, Zhang M, Wong PSJ, Li MI, Mak KW, Martin-Park A, Contreras-Perera Y, Puerta-Guardo H, Manrique-Saide P, Ng LC, Xi Z. Wolbachia wAlbB remains stable in Aedes aegypti over 15 years but exhibits genetic background-dependent variation in virus blocking. PNAS Nexus. 2022 Sep 22;1(4):pgac203. doi: 10.1093/pnasnexus/pgac203. eCollection 2022 Sep. PMID 36714832
- [Background] Lim JT, Bansal S, Chong CS, Dickens B, Ng Y, Deng L, Lee C, Tan LY, Chain G, Ma P, Sim S, Tan CH, Cook AR, Ng LC. Efficacy of Wolbachia-mediated sterility to reduce the incidence of dengue: a synthetic control study in Singapore. Lancet Microbe. 2024 May;5(5):e422-e432. doi: 10.1016/S2666-5247(23)00397-X. Epub 2024 Feb 8. PMID 38342109
- [Background] Martin-Park A, Che-Mendoza A, Contreras-Perera Y, Perez-Carrillo S, Puerta-Guardo H, Villegas-Chim J, Guillermo-May G, Medina-Barreiro A, Delfin-Gonzalez H, Mendez-Vales R, Vazquez-Narvaez S, Palacio-Vargas J, Correa-Morales F, Ayora-Talavera G, Pavia-Ruz N, Liang X, Fu P, Zhang D, Wang X, Toledo-Romani ME, Xi Z, Vazquez-Prokopec G, Manrique-Saide P. Pilot trial using mass field-releases of sterile males produced with the incompatible and sterile insect techniques as part of integrated Aedes aegypti control in Mexico. PLoS Negl Trop Dis. 2022 Apr 26;16(4):e0010324. doi: 10.1371/journal.pntd.0010324. eCollection 2022 Apr. PMID 35471983
- [Background] Zheng X, Zhang D, Li Y, Yang C, Wu Y, Liang X, Liang Y, Pan X, Hu L, Sun Q, Wang X, Wei Y, Zhu J, Qian W, Yan Z, Parker AG, Gilles JRL, Bourtzis K, Bouyer J, Tang M, Zheng B, Yu J, Liu J, Zhuang J, Hu Z, Zhang M, Gong JT, Hong XY, Zhang Z, Lin L, Liu Q, Hu Z, Wu Z, Baton LA, Hoffmann AA, Xi Z. Incompatible and sterile insect techniques combined eliminate mosquitoes. Nature. 2019 Aug;572(7767):56-61. doi: 10.1038/s41586-019-1407-9. Epub 2019 Jul 17. PMID 31316207